MBCT Delivered Via Group Videoconferencing for ACS Syndrome Patients With Depressive Symptoms

NCT04231097

April 4<sup>th</sup>, 2023

## 6. DATA ANALYSIS

6.2. Aim 2: Open pilot trial. This is a small, single-arm, pilot feasibility trial to establish preliminary feasibility and acceptability of the intervention to inform intervention adaptations for a future randomized trial. This is not a randomized clinical trial to explore efficacy of treatment on outcomes. As such the analyses are focused on descriptive statistics. Frequencies and proportions will be calculated to assess feasibility outcomes. Feasibility outcomes are: recruitment feasibility (percent of participants who consent to screening; percent of participants meeting screening criteria; percent of eligible patients who consent); MBCT feasibility (percent of participants adherent to the MBCT intervention; percent of participants retained at postintervention); videoconferencing feasibility (percent of connections dropped during sessions); and blood spot feasibility (percent of blood spot sample completion at baseline; percent of blood spot sample completion at post-intervention; percent of blood spot samples completed at followup; percent of adequate blood spot samples submitted). Means and standard deviations or medians and interquartile ranges will be calculated to assess acceptability ratings. Acceptability outcomes are rated from 0-10 with higher scores indicating greater acceptability and consist of: MBCT acceptability (helpfulness for mood; usefulness of session components); videoconferencing acceptability (ratings of videoconferencing ease of use; ratings of videoconferencing quality surveys; ratings of videoconferencing satisfaction); and blood spot acceptability (ease of blood spot collection; discomfort of blood spot collection).